CLINICAL TRIAL: NCT03867929
Title: Serum Levels of 25-Hydroxy Vitamin D in Patients With Moderate and Severe Erectile Dysfunction
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Mustafa Ozan HORSANALI, Principal investigator, Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: 2
Record Dates: First submitted 2019-02-22; First posted 2019-03-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Erectile Dysfunction
Keywords: Erectile dysfunction; Vitamin-D; Hypogonadism; Endothelial Dysfunction; Nitric Oxide
MeSH Terms: conditions — Erectile Dysfunction; Hypogonadism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 15 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- STUDY: Patient with serum 25-Hydroxy vitamin D level <27.32
  Interventions: Other: 25-Hydroxy vitamin D
- CONTROL: Patient with serum 25-Hydroxy vitamin D level >27.32
  Interventions: Other: 25-Hydroxy vitamin D

INTERVENTIONS:
Other: 25-Hydroxy vitamin D — 27.32 is calculated as a cut fo level for 25 hydroxy vitamin D deficiency

SUMMARY:
In present study, we aimed to investigate the association between erectile function severity of serum 25-Hydroxyvitamin-D and cut-off level to treat men with erectile dysfunction.

DETAILED DESCRIPTION:
Investigators retrospectively analysed 130 patients admitted to the complaint of erectile dysfunction between aged between 18-80 years old from June 2017 to October 2018 at Cigli Region Training Hospital Urology department and Recep Tayyip Erdogan University Urology Department. International index of erectile function-5 (IIEF-5) Turkish validated short form quesstionaire was performed to all patients. Antropometric characteristics including weight, height, waist circumference, body mass index (BMI) and presence of comorbide diseases were recorded. After detailed history and physical examination performed all patients, overnight fasting in the morning between 08:00-10:00, blood samples from antecubital vein were performed and serum glucose, lipid profile, follicular stimulating hormon (FSH), Luteinizing hormone (LH), total testosterone, prolactin, estradiol, 25(OH)D level were analysed. Presence of uncontrolled diabetes mellitus, uncontrolled hypertension, uncontrolled lipid metabolism disorders, neurological diseases, heamatological diseases, urinary tract infection, malignencies, chronic kidney failure, metabolic syndrome, psychiatric diseases and/or medical treatment, smoking, history of pelvic surgery, cardiac surgery and pelvic radiotherapy were accepted as exclusion criterias from the study. After IIEF-5 score adjust as 21 point, ROC analyse was used to calculate the cut-off value of 25(OH)D and level of 27.32 ng/mL was calculated as cut-off value. Patients were divided into two group according to 27.32 ng/mL level as a cut off value. Serum 25(OH)D level was lower than 27.32 ng/mL in group 1 (severe and moderate symptomatic group) and higher than 27.32 ng/mL in group 2 (mild symptomatic group).

ELIGIBILITY:
Inclusion Criteria:

* presence of erectile dysfunction

Exclusion Criteria:

* Presence of uncontrolled diabetes mellitus,
* Presence of uncontrolled hypertension,
* Presence of uncontrolled lipid metabolism disorders,
* Presence of neurological diseases,
* Presence of heamatological diseases,
* Urinary tract infection,
* Diagnosis of any malignencies,
* Chronic kidney failure,
* Presence of metabolic syndrome,
* Presence of psychiatric diseases and/or medical treatment,
* Smoking,
* History of pelvic surgery, cardiac surgery and pelvic radiotherapy

Ages: 18 Years to 80 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes — erectile dysfunction
Study Population: patients with erectile dysfunction aged between 18 and 80 years
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Laboratory results | 1 year
  Serum 25 Hydroxy vitamin D levels (ng/mL), group 1 include patients with serum 25 hydroxy vitamin D levels higher than 27.32 ng/ml and Group 2 include patients with serum 25 hydroxy vitamin D levels lower than 27.32 ng/mL
Clinical results | 1 year
  IIEF-5 quesstionaire score (0-15 point is severe erectile dysfunction, 16-21 point is moderate erectile dysfunction and >21 point is mild erectile dysfunction)

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Ozan Horsanalı, Dr., Principal Investigator — Cigli Regional Training Hospital, Urology Department
Locations (1):
- Cigli Regional Training Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No